CLINICAL TRIAL: NCT02700581
Title: Impact of Moderate Positive End-expiratory Pressure on Hepatic Venous Flow in Patients Undergoing Cardiac Surgery
Brief Title: Impact of Positive End-expiratory Pressure on Hepatic Venous Flow
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, Professor of Anesthesiology, Konkuk University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KUH000000 TBD
Record Dates: First submitted 2016-02-23; First posted 2016-03-07 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Valvular Heart Disease
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- low PEEP conventional ventilation (Active Comparator): PEEP 2 mmHg tidal volume 10ml/kg
  Interventions: Procedure: low PEEP conventional ventilation
- moderate PEEP conventional ventilation (Experimental): PEEP 7 mmHg tidal volume 10ml/kg
  Interventions: Procedure: moderate PEEP conventional ventilation
- low PEEP protective ventilation (Experimental): PEEP 2 mmHg with tidal volume 6 ml/kg
  Interventions: Procedure: low PEEP protective ventilation
- moderate PEEP protective ventilation (Experimental): PEEP 7 mmHg tidal volume 6ml/kg
  Interventions: Procedure: moderate PEEP protective ventilation

INTERVENTIONS:
Procedure: low PEEP conventional ventilation
  Arms: low PEEP conventional ventilation
Procedure: moderate PEEP conventional ventilation
  Arms: moderate PEEP conventional ventilation
Procedure: low PEEP protective ventilation
  Arms: low PEEP protective ventilation
Procedure: moderate PEEP protective ventilation
  Arms: moderate PEEP protective ventilation

SUMMARY:
The purpose of this study is to determine the difference in the impact of moderate positive end-expiratory pressure (PEEP) on hepatic venous flow Doppler in patients undergoing cardiac surgery: conventional versus protective ventilation strategy The possible changes in forward and backward flows (Doppler profiles) of hepatic venous flow at different degrees of PEEP in conventional and protective ventilation strategies are analyzed by using intraoperative transesophageal echocardiography (TEE) in patients undergoing cardiac surgery .

DETAILED DESCRIPTION:
Following data would be determined after 5 min-exposure volume controlled ventilation employing tidal volume of 10 ml/kg and 6 ml/kg with low PEEP (with 2 mmHg) and moderate PEEP (7 mmHg) during remifentanil-based anesthesia (1.0 mcg/kg/min) for cardiac surgery (n=12)

1. sum of forward hepatic venous flow
2. sum of backward hepatic venous flow
3. peak velocity of diastolic hepatic venous flow
4. lung compliance
5. peak airway pressure
6. mean airway pressure
7. other pressure derived hemodynamic parameters:heart rate; systolic, diastolic, and mean blood pressures; systolic, diastolic, and mean pulmonary artery pressures; central venous pressure (CVP), pulmonary capillary

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery
* Patients provide written informed consents

Exclusion Criteria:

* Re-do or tri-do surgery
* Patients with active infection
* Patients with endocrine disease
* Patients ischemic heart disease
* patients with tricuspid valve regurgitation greater than mild degree

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-04 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
forward hepatic venous flow | 3 min after intervention
  Hepatic venous flow Doppler, cm/sec, by transesophageal echocardiography

SECONDARY OUTCOMES:
reversed hepatic venous flow | 3 min after intervention
  Reversed hepatic venous flow Doppler, cm/sec, by transesophageal echocardiography

IPD SHARING:
Plan to Share IPD: No